CLINICAL TRIAL: NCT01175538
Title: Primary Prophylaxis of Hepatic Encephalopathy in Patients With Cirrhosis: an Open Labeled Randomized Controlled Trial of Lactulose Versus no Lactulose
Brief Title: Primary Prophylaxis of Hepatic Encephalopathy in Patients With Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Prof Barjesh Chander Sharma, G B Pant Hospital
Purpose: Treatment
Other Study IDs: PS001
Record Dates: First submitted 2010-08-02; First posted 2010-08-05 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2009-10

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic encephalopathy; Lactulose
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lactulose (Experimental)
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Lactulose — In the Gp-L group, patients will receive 30-60 ml of lactulose in 2 or 3 divided doses so that patient passes 2-3 semisoft stools per day
Drug: Lactulose — lactulose will be used in 30-60ml/day

SUMMARY:
To assess the effects of lactulose for the prevention of first episode of altered sensorium (hepatic encephalopathy, primary prophylaxis) in patients with cirrhosis.

DETAILED DESCRIPTION:
Development of hepatic encephalopathy in a patient with cirrhosis is associated with poor survival rate of 10-70% at one year depending upon hepatic and renal functions. Treating patients to prevent development of first episode of hepatic encephalopathy is classified as primary prophylaxis of hepatic encephalopathy and preventing recurrence of hepatic encephalopathy in patients who had previous episode of hepatic encephalopathy is secondary prophylaxis of hepatic encephalopathy

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic patients(18-70yrs) who never had encephalopathy

Exclusion Criteria:

* history of taking lactulose in the past 6 weeks
* alcohol intake during the past 6 weeks
* hepatocellular carcinoma
* previous TIPS or shunt surgery
* significant co morbid illness such as heart, respiratory, or renal failure
* neurologic diseases such as alzheimer's disease, parkinson's disease and nonhepatic metabolic encephalopathies.
* patients on psychoactive drugs such as antidepressants or sedatives
* who restarted alcohol during follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
prevention of first episode of hepatic encephalopathy | 6 months

SECONDARY OUTCOMES:
Side effects to lactulose and mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Barjesh C Sharma, MD,DM, Principal Investigator — G B Pant Hospital New Delhi 110002
Locations (1):
- G B Pant Hospital, New Delhi, National Capital Territory of Delhi, India